CLINICAL TRIAL: NCT05358041
Title: Comparing Diagnostic Yield of Real Time Cone Beam Computer Tomography Guided Electromagnetic Navigational Bronchoscopy With Cone Beam Computer Tomography Guided Robotic Navigational Bronchoscopy for Peripheral and Central Lung Lesions
Brief Title: Cone Beam CT Guided Robotic Navigational Bronchoscopy
Acronym: CBCTRNB
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Columbus Regional Health (Other)
Responsible Party: Principal Investigator, Deepankar Sharma, Medical Director, Lung Institute and Section Chief, Pulmonary & Critical Care, Columbus Regional Health
Other Study IDs: 007
Record Dates: First submitted 2022-04-26; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Lung Nodule; Lung Mass; Lung Cancer
Keywords: Lung Nodule; Lung Mass; Lung Lesion; Cone Beam CT CT Augmented Fluoroscopy; Electromagnetic Navigation Bronchoscopy; Robotic Navigation Bronchoscopy; Shape Sensing Navigational Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electromagnetic Navigational Fixed Angle Bronchoscopy with CBCT Guidance: Patient is undergoing electromagnetic navigation bronchoscopy using Medtronic super D version 7 EMN system, peripheral endobronchial ultrasound and Cone Beam CT Guidance using the Philips Azurion 7 C20 FlexMove with Embo Guide and Overlay software to create CT Augmented Fluoroscopy under general anesthesia.
- Robotic Shape Sensing Bronchoscopy with CBCT Guidance: Patient is undergoing robotic navigation bronchoscopy using IOn robotic platform, peripheral endobronchial ultrasound and Cone Beam CT Guidance using the Philips Azurion 7 C20 FlexMove with Embo Guide and Overlay software to create CT Augmented Fluoroscopy under general anesthesia.
  Interventions: Device: Robotic Bronchoscopy

INTERVENTIONS:
Device: Robotic Bronchoscopy — Replace the Super-D EMN navigational platform with Ion Robotic bronchoscopy platform guided with shape sensing technology
  Groups: Robotic Shape Sensing Bronchoscopy with CBCT Guidance

SUMMARY:
Navigational bronchoscopy (NB) is used to access peripheral and central parenchymal lung lesions via endobronchial and transbronchial approach. Currently there are multiple platforms available to provide guidance to reach the peripheral and central lesions in the lung which are inaccessible via traditional video bronchoscopy. Traditionally NB is done under fluoroscopic guidance using C-arm but with development of Cone Beam CT and 3D reconstruction technology, fluoroscopy can be enhanced to much higher resolution and can also provide real time 3D augmentation of the lesion. It also enables the user to obtain a CT of the Chest to confirm the real time location of the lesion and the bronchoscopic biopsy catheter and instruments. This has proven to improve the yield and sensitivity of Navigational bronchoscopic guided Biopsy of the lung nodules and masses. Out of the various navigational platforms we have, most of them are based on Electromagnetic guidance and some on Shape sensing technology. Some of the platforms have fixed angle catheter while the newer robotic platforms have articulating catheters with much more range of motion. So far we do not have any data directly comparing the diagnostic yield of Electromagnetic navigational bronchoscopy with Robotic shape sensing guided bronchoscopy while using Cone Beam CT and Augmented fluoroscopy with both the platforms. With my study, I want to examine the change in diagnostic yield and sensitivity of fixed angle ENB guided bronchoscopy and articulating robotic shape sensing bronchoscopy both using Cone Beam CT with 3D reconstruction.

DETAILED DESCRIPTION:
Navigation bronchoscopy (NB) has been used for more than a decade to access peripheral and central parenchymal lung lesions bronchoscopically. Traditionally standard fluoroscopy using C-arm is used to confirm the location and guide the biopsy instruments under real-time guidance. With availability of Cone Beam CT, fluoroscopic images of much higher quality and resolution can be obtained intra-operatively. It also enables the bronchoscopist to obtain intraoperative CT images and confirm the exact location of the lesion and the Bronchoscopic biopsy catheter or the biopsy instruments.

Recently we have had significant advancements in the technology to guide and operate the instruments used to reach these hard to reach lesions within the lungs. We have different fixed angle electromagnetic guided platforms, articulating robotic electromagnetic guided platforms and articulating robotic shape sensing guided platforms.

At my institution, lung nodules/masses requiring NB has evolved over the years starting from Medtronic Super-Dimension Version 7 Electromagnetic Navigational Bronchoscopy (ENB) system to ION Robotic Bronchoscopy platform (RNB). All the procedures are done under fluroscopic guidance which has also evolved from a regular C-Arm to Philips Cone Beam CT with Augmented Fluoroscopy.

During this evolution we have had Medtronic Super-D ENB with 2D fluoro followed by Medtronic Super-D ENB with CBCT and Augmented fluoroscopy and now have the Ion robotic platform with CBCT and Augmented fluoroscopy with low dose protocol.

All the lesions are confirmed using peripheral/radial Endobronchial Ultrasound (rEBUS). Once the appropriate location is reached, biopsy is obtained using FNA (18G or 21G), Single or Triple needle brush, Transbronchial forceps and Bronchoalveolar lavage is done for cytology or micro studies if needed.

A pathologist is present on site for all the cases to review the slides and assist in diagnosis. All the cases are done under general anesthesia through endotracheal tube.

Also, all the NB procedures have been performed by one Interventional Pulmonologist since August 2017.

For the interventional arm, all the aspects will remain the same except that the procedure will utilize Ion Robotic bronchoscopy platform and pre-operatively every patient will undergo incentive spirometry, dual short acting bronchodilator treatment and will be maintained at relatively higher PEEP and Lower FiO2 than before.

The diagnostic yield will be compared to the patients who underwent procedure using Super-D Electromagnetic platform with CBCT and Augmented Fluoroscopy.

All cases are still done in Hybrid ORand all the patients are completely paralyzed intra-operatively. Also, all procedures in both arms will use a Philips Azurion 7 C20 FlexMove system with Emboguide, 3D Segmentaion and Overlay tools. This enables the bronchoscopist to obtain a CT scan of the chest and also segment out the lesion(s) of interest and to overlap the 3-D image of the lesion on live fluoroscopy in all 3 dimensions.

During the ENB and RNB procedures, at least 1 full Xpert CT is obtained, mostly after completing the airway registration and advancing the guided catheter to the lesion of interest. Once the extended working channel and the locatable guide or The robotic articulating catheter is advanced to the lesion using ENB/Shape sensing guidance, the catheter is held at that position and patient is maintained in inspiratory breath hold and Cone Beam CT is used to obtain the Xpert CT that shows the lesion and surrounding lungs, chest and mediastinal structures in the surrounding area of the chest. This is then used to analyze the location of the lesion and the lesion of the extended working channel/robotic catheter and the biopsy instruments in relation to the lesion. The lesion is then segmented and EmboGuide + Overlay feature is used to project a 3D view of the lesion on the live fluoroscopic images in all three axis. This also allows the bronchoscopist to obtain Anterior-posterior, Lateral and oblique views at various angles while maintaining the 3D overlap.

Additional CT scans might be obtained intra-operatively if needed to guide the biopsy catheter appropriately towards the lesion.

Due to the live nature of the Cone Beam CT, it is much more capable of providing accurate guidance regarding the location of the lesion and the biopsy instruments. hence, in case of any discrepancy, information provided by Cone Beam CT is considered more reliable and used with higher confidence.

Rest of the steps involved in procedure are similar between the control and the interventional arm including the surgeon, type of biopsy instruments, use of peripheral Endobronchial Ultrasound and availability of on-site pathologist. The biopsy instruments include transbronchial needle for FNA, Single or triple needle brush and transbronchial forceps. Bronchoalveolar lavage is also obtained at the end via working channel.

All the patients undergoing biopsy of the peripheral/central lung lesions using ENB/RNB also undergo Convex EBUS guided mediastinal surveillance and EBUS-TBFNA of any Lymph Node that appears to be greater than 5 mm on EBUS exam.

My study aims to study the difference in diagnostic yield and sensitivity of electromagnetic navigational bronchoscopy with fixed angle catheter vs robotic shape sensing bronchoscopy with articulating catheter while using Cone Beam CT with segmentation, 3-D overlay and CT augmented fluoroscopy for diagnosis of peripheral and central lung lesions including lung nodules and masses which could not be directly accessed using just white light bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung nodule
* Patients with lung mass
* Patients undergoing navigation bronchoscopy for biopsy of peripheral/central lung lesions.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients unable to complete the navigational bronchoscopy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodule, mass or lesion undergoing navigation bronchoscopy for biopsy. Majority of the patients are smokers. Some of the patients are found to have the lung nodule, mass or lesion incidentally or on the low-dose CT for lung cancer screening.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2022-11-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for malignancy | 1 year
  Percentage of malignant lesions accurately diagnosed on biopsy
Diagnostic Yield | 1 year
  Percentage of correct underlying diagnosis

SECONDARY OUTCOMES:
Procedural Complications | 1 year
  Pneumothorax or Bleeding
Intra-Operative time | 1 year
Radiation Exposure | 1 year
  Will have a record of radiation dose from the Cone Beam CT data for both the arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbus Regional Health, Columbus, Indiana, United States

IPD SHARING:
Plan to Share IPD: No